CLINICAL TRIAL: NCT04709380
Title: Phase III Randomized Clinical Trial of Radiotherapy Plus Toripalimab Versus Sorafenib in Advanced Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis
Brief Title: Phase III RCT of Radiotherapy Plus Toripalimab Versus Sorafenib in Advanced Hepatocellular Carcinoma With PVTT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: IDMC recommended to terminate the study since Interim analysis showed that the experimental group had significant superiority over the control group in TTP and OS (p<0.001), meeting the predefined interim analysis endpoints in the study protocol.
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, BO CHEN, Associate Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2509
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Radiotherapy; Toripalimab; Sorafenib; Advanced Hepatocellular Carcinoma
Keywords: Radiotherpay; Anti-PD-1 antibody; Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — Radiotherapy; toripalimab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy plus Toripalimab (Experimental): Patients in the experimental group will be given local vein tumor thrombus/hepatic vein tumor thrombus +/- intrahepatic large lesions with hypofractionated intensity modulated radiotherapy (tumor area dose 40-60Gy/10-20f), concurrent with and followed by 240mg Q3W of toripalimab within 1 week of radiotherapy.
  Interventions: Other: Radiotherapy plus Toripalimab
- Sorafenib (Active Comparator): Patients in the control group will be treated with sorafenib (400mg, twice a day).
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Other: Radiotherapy plus Toripalimab — Intensity modulated radiotherapy has shown important role in the treatment of hepatocellular carcinoma (HCC), especially for advanced disease with portal vein tumor thrombosis (PVTT), or hepatic vein tumor thrombosis. Toripalimab is a recombinant, humanized programmed death receptor-1 (PD-1) monoclonal antibody that binds to PD-1 and prevents binding of PD-1 with programmed death ligands 1 (PD-L1) and 2 (PD-L2).
  Arms: Radiotherapy plus Toripalimab
Drug: Sorafenib — Sorafenib is a multi-targeted oral drug for the treatment of cancer.Treatment of inoperable advanced renal cell carcinoma ,inoperable or distant metastatic primary hepatocellular carcinoma and so on.
  Arms: Sorafenib

SUMMARY:
To explore the efficacy of radiotherapy plus toripalimab Versus standard treatment of sorafenib in advanced hepatocellular carcinoma with Portal Vein/Hepatic vein Tumor Thrombosis.

DETAILED DESCRIPTION:
This is an single-center, open, randomized study, which is going to enroll patients filtered to meet the standard of advanced hepatocellular carcinoma, in a 2: 1-proportional randomly assigned to the test group and control group. Patients in the experimental group will be given local vein tumor thrombus/hepatic vein tumor thrombus +/- intrahepatic large lesions with hypofractionated intensity-modulated radiotherapy (tumor area dose 40-60Gy/10-20f), concurrent with and followed by 240mg Q3W of toripalimab within 1 week of radiotherapy started. Patients in the control group will be treated with sorafenib (400mg, twice a day).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical or histologic diagnosis of Hepatocellular carcinoma (HCC) according to the 2019 version of liver cancer diagnosis and treatment guideline.
2. Aged between 18 and 80 years.
3. ECOG 0-1.
4. The left volume of liver-GTV which is received less than dose of 5Gy is more than 250ml after the portal vein/hepatic vein tumor thrombosis and its connected primary main lesion is received treatment dose of 40-60Gy/10-20f.
5. Patients may have a history of treatments for hepatocellular carcinoma such as TACE, radiofrequency, surgery, chemotherapy, and Chinese herbal medicine, but all patients must have not been received targeted therapy and Immunotherapy, such as anti-PD-1, anti-PD-L1 or anti-PD-L2 drug therapy.
6. BCLC Stage C, HCC combined with portal vein or hepatic vein tumor thrombosis. If it is a portal vein tumor thrombosis, it must involve the left or right portal trunk at least. If it is a hepatic vein tumor thrombosis, it must involve the left or middle or right main hepatic veins at least. At the same time, eligible patients have to meet one of the following conditions. (1) There are distant metastases (except for central nervous system and meningeal metastases); (2) Both hepatic lobes are showed multiple lesions which are unable to be fully covered within the target area; (3) portal vein tumor thrombosis involved main portal trunk.
7. The expected lifetime is more than 3 months.
8. Child A5, A6, B7.
9. Virus conditions: HBV DNA <2000 IU/mL, if ≥ 2000 IU/mL, need to accept antiviral treatment until<2000 IU/mL; patients with a positive HCV antibody must have a negative polymerase chain reaction (PCR) test result of HCV RNA;
10. Liver function: ALT is within 2.5 times of the upper limit of normal. AST can be within 6 times of the upper limit of normal if ALT is within 1.5 times of the upper limit of normal and cardiac infarction is excluded. If ALT is 1.5 to 2.5 times the upper limit of normal, AST must be within 1.5 times the upper limit of normal.
11. There is no obvious abnormality in the electrocardiography, and no obvious cardiac dysfunction.
12. Renal function: CRE and BUN are within 1.5 times the upper limit of normal.
13. Blood routine test: Hb≥80g/L, ANC≥1.0×10 9/L, PLT≥40×10 9/L.
14. Coagulation function: no bleeding tendency.
15. Willingness to voluntarily participate in the clinical trial and sign informed consent..

Exclusion Criteria:

1. Those who are participating in other clinical trials.
2. Had prior abdominal irradiation, or had prior liver transplantation.
3. Patients with chronic, serious diseases such as cardiac, pulmonary, and renal disease.
4. Suspected or true alcohol, drug abuse history.
5. May be allergic to treatment with sorafenib or toripalimab.
6. Have received immunotherapy in the past, such as anti-PD-1, anti-PD-L1, anti-PD-L2 drugs, and other drugs that stimulate or co-inhibitory T cell receptors (such as CTLA-4, OX- 40 or CD137) treatment
7. Severe mental or nervous system disorders that affect informed consent and/or expression or perception of adverse events.
8. Previous clinical diagnosis of hepatic encephalopathy in the past 6 months. Patients with hepatic encephalopathy which are controlled by rifaximin or lactulose are not allowed to participate in the study.
9. Moderate to severe ascitic fluid with obvious symptoms.
10. Concomitant secondary malignant tumors or other tumors (except superficial skin cancer, localized low-grade malignant tumors and carcinoma in situ) within 3 years before the start of the study.
11. History of gastrointestinal hemorrhage within 6 months before the start of the study, or was diagnosed by ERCP/CT/DSA as a high risk of rupture and bleeding of esophageal gastric varices.
12. Suffer from serious unhealed wounds, ulcers or fractures.
13. Active central nervous system metastasis or cancerous meningitis.
14. Active tuberculosis (TB), who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before the first medication.
15. History of biliary fistula, gastrointestinal perforation, and intra-abdominal abscess within 4 weeks before the start of the study.
16. History of unstable angina, myocardial infarction, coronary artery bypass grafting, congestive heart failure, cerebrovascular accident (including transient ischemic attack, pulmonary embolism) within 3 months before the start of the study.
17. NCI-CTCAE v.4 grade ≥2 cardiac arrhythmia, atrial fibrillation, or QT interval prolongation of any NCI-CTCAE v.4 grade (male > 450ms, female > 470ms).
18. Uncontrollable hypertension treated with best antihypertensive drugs (> 150/90mmHg after rational medication).
19. History of HIV infection.
20. Females who are pregnant or breastfeeding.
21. Live vaccines were vaccinated within 30 days before the first dose of study drug. Live vaccines include but are not limited to the following: measles, mumps, rubella, varicella/shingles (chickenpox), yellow fever, rabies, BCG (BCG) and typhoid vaccines. Since seasonal influenza vaccines for injection are usually inactivated virus vaccines, their use is allowed; however, intranasal influenza vaccines (for example, FluMist) are live attenuated vaccines, so they are not allowed.
22. Have an active autoimmune disease that requires systemic treatment in the past 2 years (for example, immunomodulatory drugs, corticosteroids, or immunosuppressive drugs. Autoimmune diseases such as autoimmune hepatitis, interstitial pneumonia, uveal Inflammation, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome related vascular thrombosis, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, Glomerulonephritis, etc., hyperthyroidism or hypothyroidism, asthma that requires bronchodilator treatment, etc.). Replacement therapy (for example, thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered systemic therapy and is allowed.
23. Combined with medical contraindications that cannot accept any contrast-enhanced imaging examinations (CT or MRI).
24. Severely allergic to research intervention and/or any of its excipients (≥Grade 3).
25. Uncontrolled metabolic disorders or other non-malignant tumor organs or systemic diseases or cancer secondary reactions, which can lead to higher medical risks and/or uncertainty in survival evaluation.
26. Patients who have received allogeneic tissue/solid organ transplantation.
27. Patients with other acute or chronic diseases, mental illnesses, or abnormal laboratory test values that may cause the following results: increase the risk related to study participation or study drug administration, or interfere with the interpretation of the study results, and the patients shall be treated according to the judgment of the investigator classified as not eligible to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
TTP | up to 24 months
  Time to Progression (TTP) was defined as the duration from the date of patient recruited to the first progress at any site or the date of death.

SECONDARY OUTCOMES:
ORR | up to 24 months
  Overall Response Rate (ORR) was defined as the total of CR (Complete Response) and PR (Partial Response). CR and PR were assessed by independent reviewers according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
OS | up to 24 months
  Overall Survival (OS) was defined as the duration from the date of patient recruited to the date of death with any reason.
Incidence of grade 3 and above adverse events | up to 24 months
  Adverse events was evaluated during received protocol therapy according to CTCAE 4.03.

CONTACTS AND LOCATIONS:
Locations (1):
- Bo Chen, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No